CLINICAL TRIAL: NCT05214469
Title: Evaluatıon of Nutrıtıonal Status and Total Antıoxıdant Capacıty in Individuals Diagnosed of Osteoarthritis
Brief Title: Evaluatıon of Nutrıtıonal Status and Total Antıoxıdant Capacıty in Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Beda Büşra ÖZALP, Principal investigator, Akdeniz University
Other Study IDs: OSTEOBEDA
Record Dates: First submitted 2021-12-15; First posted 2022-01-28 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis; Knee Osteoarthritis; Antioxidant Capacity; Oxidant Capacity; Nutrition
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case Group: Individuals diagnosed with knee-osteoarthritis
- Control Group: Individuals who do not have a chronic disease and are not diagnosed with osteoarthritis

SUMMARY:
This is a descriptive cross-sectional study conducted to evaluate the nutritional status and total antioxidant/oxidant capacity of individuals diagnosed with osteoarthritis.

DETAILED DESCRIPTION:
The aim of this study is to determine the nutritional status of individuals diagnosed with osteoarthritis, to evaluate dietary total antioxidant/oxidant capacity and serum total antioxidant/oxidant capacity, and to examine the relationship of total antioxidant capacity with anthropometric measurements and nutritional status.

The study will include adult individuals diagnosed with osteoarthritis who applied to the Physical Therapy and Rehabilitation polyclinics of Ankara City Hospital. After the individuals fill out the questionnaire containing information about their socio-demographic characteristics, nutritional habits and physical activity levels, the researchers will take the food consumption records and the frequency of food consumption with a 24-hour reminder method. The total antioxidant amount of the diet will be determined from the food consumption records of the individuals. In addition to these, anthropometric measurements of individuals such as height, body weight and waist circumference will also be taken by the researchers.

In the study, routine biochemical parameter will be recorded from patient files and serum total antioxidant/oxidant capacity values will be examined.

The sample calculation was made using the Vanderbilt University Sample Calculation Tool, benefiting from the antioxidant capacity researches previously done in individuals with osteoarthritis in the literature. Assuming a standard deviation of ±20 in the study, the minimum sample size to be taken with 80% power and 5% error was determined as at least 47 people (case group) and 30 people (control group). In terms of the correct interpretation of the research results, the individuals in the case and control groups were similar in terms of age, gender and BMI in the selection of the sample (p≥0.05).

In the study, descriptive statistics (mean, lower value, upper value, standard deviation, standard deviation, mean) for data such as anthropometric measurements, daily consumption of food groups, energy and nutrient intakes, food consumption amounts and the rate of meeting the needs of energy and nutrients (%), number of meals. median) was calculated. The conformity of the variables to the normal distribution was examined using the Shapiro-Wilk test. Student's t test was used for the comparison of normally distributed variables in the groups (osteoarthritis diagnosis-control group), and the Mann-Whitney-U test was used for the comparison of non-normally distributed variables. In the comparison of more than two measurements, the Friedman test was used in cases where the normal distribution was not suitable. Correlations between numerical data were evaluated with the Pearson correlation test. The analyzes of the study were made in the SPSS 22.0 statistical package program and the statistical significance level was accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65,
* Being followed up with a diagnosis of knee-osteoarthritis by doctor

Exclusion Criteria:

* Individuals under 18 and over 65 years of age,
* Individuals with acute or chronic inflammatory diseases,
* Individuals with chronic diseases,
* Individuals who consume alcohol,
* Smokers,
* Individuals who have not taken additional vitamin and mineral supplements in the last 6 months,
* Individualswho are not volunteer to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outpatient clinic patients
Sampling Method: Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Total Antioxidant and Oxidant Capacity | Blood samples will be obtained once on the first day after inclusion. Samples will be stored in -80 C medical refrigerator and analysis will be done after collection of all samples.
  Higher total antioxidant capacity is better and higher oxidant capacity is worse.
Dietary Total Antioxidant Capacity | Will be obtained only once on the first day after inclusion.
  In order to evaluate the food consumption of the individuals, the food consumption frequency form (with their amounts) will also be applied. The dietary total antioxidant capacity (TAC) will be estimated using a FRAP (ferric reducing antioxidant potential).

SECONDARY OUTCOMES:
Osteoarthritis Stage | Will be obtained only once on the first day before inclusion.
  Bilateral knee radiographs taken at the diagnosis stage will be interpreted by the doctor according to the Kellgren Lawrence staging system and osteoarthritis staging will be recorded. Osteoarthritis is deemed present at grade 2 although of minimal severity. Each radiograph will be assigned a grade from 0 to 4, which they correlated to increasing severity of OA, with Grade 0 signifying no presence of OA and Grade 4 signifying severe OA.
Physical Activity Status | Will be done obtained only once on the first day after inclusion.
  To determine the physical activity status of the participants. International Physical Activity Questionnaire-Short Form will be applied. Form will be applied and used to assess their physical condition. Higher score means more energy expended carrying out physical activity.
Height Measuring | Will be done obtained only once on the first day after inclusion.
  The height will be made with the height measuring tool of the scale.The head is level with a horizontal Frankfurt plane (below - an imaginary line from the lower border of the eye orbit to the auditory meatus).
Weight Measuring | Will be done obtained only once on the first day after inclusion.
  The body weights of the individuals participating in the research will be measured with a precision scale (±0.1 kg sensitive) that is calibrated at regular intervals, without shoes and wearing as light clothes as possible.
Body Mass Index (BMI) | Will be done obtained only once on the first day after inclusion.
  Body Mass Index (BMI), which is very important in the detection and evaluation of obesity or malnutrition; It will be calculated as kg/m² with the formula of body weight/height.

CONTACTS AND LOCATIONS:
Overall Officials: Nilgün SEREMET KÜRKLÜ, Asist. Prof., Study Director — Akdeniz University, Faculty of Health Sciences, Nutrition and Dietetics, Antalya, TURKEY; Beda ÖZALP, Dietetican, Principal Investigator — Akdeniz University, Faculty of Health Sciences, Nutrition and Dietetics, Antalya, Turkey; Emre ADIGÜZEL, Assoc. Prof., Study Chair — Ankara City Hospital, Physical Medicine and Rehabilitation Hospital, Ankara, TURKEY; Kübra Tel Adıgüzel, Asist. Prof., Study Chair — University of Health Sciences, Faculty of Health Sciences, Nutrition and Dietetics, Ankara, TURKEY
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)